CLINICAL TRIAL: NCT00782379
Title: A Phase II Trial of Myeloablative Conditioning and Transplantation of Partially HLA-Mismatched Peripheral Blood Stem Cells for Patients With Hematologic Malignancies
Brief Title: Combination Chemotherapy, Donor Stem Cell Transplant, Tacrolimus, Mycophenolate Mofetil, and Cyclophosphamide in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northside Hospital, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000617648; BMTGG-NSH-864
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-03

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes
Keywords: stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic | interventions — Busulfan; Cyclophosphamide; fludarabine phosphate; Mycophenolic Acid; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myeloablative Haploidentical Transplant (Experimental): All patients will receive treatment using Fludarabine, Busulfan and Cyclophosphamide prior to receiving a haploidentical transplant followed by post-transplant cyclosphosphamide.
  Interventions: Drug: busulfan; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Drug: tacrolimus; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Drug: busulfan — 110 mg/m2 infused over 3 hours once daily on 4 consecutive days (Days -7, -6, -5, -4)
Drug: cyclophosphamide — 14.5 mg/kg infused over 1-2 hours once daily on 2 consecutive days (days -3,-2).
Drug: fludarabine phosphate — 30mg/m2 infused over 30 minutes once daily on three consecutive days (days -5, -4, -3)
Drug: mycophenolate mofetil — 15 mg/kg po three times a daily with a maximum dose of 3gm/day starting D+5. To be discontinued on Day +35 in the absence of clinically significant GVHD.
  Other Names: CellCept
Drug: tacrolimus — 0.03 mg/kg/day infuse over 24 hours starting on day +5 (adjusted to maintain trough level of 5-15 ng/ml). Switch to oral (twice daily divided dose) on day +21 or when able to tolerate PO. Discontinue on day +180 in the absence of clinically significant GVHD.
  Other Names: Prograf, FK-506
Procedure: allogeneic hematopoietic stem cell transplantation — Patients to received unmanipulated PBSCs on Day 0
  Other Names: Allo HSCT
Procedure: peripheral blood stem cell transplantation — patients to receive unmanipulated PBSCs on day 0
  Other Names: allogeneic hematopoietic stem cell transplant

SUMMARY:
RATIONALE: Giving chemotherapy, such as fludarabine, busulfan, and cyclophosphamide, before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving high-dose cyclophosphamide together with tacrolimus and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well combination chemotherapy works when given together with a donor stem cell transplant, followed by tacrolimus, mycophenolate mofetil, and high-dose cyclophosphamide, in treating patients with high-risk hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the incidence of graft rejection and severe graft-versus-host disease after myeloablative HLA-mismatched peripheral blood stem cell transplantation (PBSCT) from first-degree relatives in patients with high-risk hematologic malignancies.

Secondary

* To estimate overall survival, relapse, non-relapse mortality, and event-free survival in these patients.
* To characterize additional hematologic and non-hematologic toxicities of myeloablative haploidentical PBSCT.
* To characterize donor hematopoietic chimerism in peripheral blood stem cells after PBSCT.

OUTLINE:

* Preparative regimen: Patients receive fludarabine phosphate IV over 30 minutes on days -7 to -2, busulfan IV over 3 hours on days -7 to -4, and cyclophosphamide IV over 1-2 hours on days -3 and -2.
* Allogeneic peripheral blood stem cell transplantation (PBSCT): Patients undergo infusion of unmanipulated peripheral blood stem cells on day 0.
* Post-transplant regimen: Patients receive high-dose cyclophosphamide IV over 1-2 hours on days 3 and 4, tacrolimus IV over 24 hours or orally twice daily on days 5-180, and oral mycophenolate mofetil 3 times daily on days 5-34 followed by a taper to day 90. Treatment continues in the absence of disease progression or clinically significant graft-vs-host disease.

After completion of PBSCT, patients are followed periodically for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following high-risk hematologic malignancies:

  * Chronic myelogenous leukemia meeting one of the following criteria:

    * Disease in chronic phase and resistant to available tyrosine kinase inhibitors
    * Disease in accelerated phase
    * Disease with blast crisis that has entered into a second chronic phase after induction chemotherapy
  * Acute myelogenous leukemia meeting the following criteria:

    * Marrow blasts < 5% but persistence of minimal residual disease by flow cytometry, cytogenetics, or FISH
    * Must meet one of the following criteria:

      * Disease in second or subsequent complete remission
      * Primary induction chemotherapy failure with disease subsequently entering complete remission
      * Disease in first complete remission with poor-risk cytogenetics or arising from preceding hematological disease
  * Myelodysplastic syndrome meeting at least one of the following criteria:

    * Treatment-related
    * Monosomy 7 or complex cytogenetics
    * International prognostic scoring system score ≥ 1.5
    * Chronic myelomonocytic leukemia
  * Acute lymphocytic leukemia or lymphoblastic lymphoma meeting the following criteria:

    * Marrow blasts < 5% but persistence of minimal residual disease by flow cytometry, cytogenetics, or FISH
    * Must meet one of the following criteria:

      * Disease in second or subsequent complete remission
      * Acute lymphocytic leukemia with poor-risk karyotype [e.g., t(9;22) or bcr-abl fusion, t(4;11), or other MLL translocation] and in first complete remission
  * Chronic lymphocytic leukemia or prolymphocytic leukemia meeting both of the following criteria:

    * Previously treated disease that has either relapsed or failed to respond adequately to conventional-dose therapy including purine analogs
    * In the opinion of the transplant physician, unlikely to benefit from reduced intensity transplantation due to the presence of one or more high-risk features (i.e., bulky tumor masses, B symptoms, and/or inadequate response to salvage chemotherapy)
  * Hodgkin or non-Hodgkin lymphoma (including low-grade, mantle cell, and intermediate-grade/diffuse disease) meeting the following criteria:

    * Previously treated disease that has either relapsed or failed to respond adequately to conventional-dose therapy or autologous transplantation
    * In the opinion of the transplant physician, unlikely to benefit from reduced intensity transplantation due to the presence of one or more high-risk features (i.e., bulky tumor masses, B symptoms, and/or inadequate response to salvage chemotherapy) NOTE: A new classification scheme for adult non-Hodgkin lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.
* No available matched related or unrelated donor OR a matched related or unrelated donor will not be available in the time frame necessary to perform a transplant
* Availability of a first-degree relative (parent, child, sibling) matched at 3/6-5/6 loci (HLA-A, -B, -DR)

  * Donor must be willing to donate mobilized peripheral blood stem cells
  * No positive HLA crossmatch in the host-vs-graft direction or high titer donor-specific antibodies

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Bilirubin < 2 mg/dL (unless due to hemolysis, Gilbert syndrome, or primary malignancy)
* Creatinine < 2 mg/dL OR creatinine clearance ≥ 40 mL/min
* Not pregnant
* Fertile patients must use effective contraception
* LVEF (Left ventriculr ejection fraction) ≥ 45%
* FEV_1 and forced vital capacity ≥ 50% predicted
* No HIV positivity
* No debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment and follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No immunosuppressive agents ≤ 24 hours after completion of post-transplant cyclophosphamide (including steroids as antiemetics)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-10; Primary Completion 2011-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R. Solomon, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia; H. Kent Holland, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia; Asad Bashey, MD, PhD, Principal Investigator — Blood and Marrow Transplant Group of Georgia; Lawrence E. Morris, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (1):
- Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were consented between 12/17/08 through 01/13/11. The transplants occured between 1/13/09 and 3/2/11
Pre-assignment Details: NA - this study did not use group assignments. All patients received the same preparative regimen consisting of Fludarabine 25 mg/m2 x 5 days, busulfan 110 mg/m2 x4 days, cyclophosphamide 14.5 mg x 2 days PRE transplant and cyclophosphamide 50 mg x2 days POST transplant
Groups:
- Haploidentical Transplant: Patients receiving Fludarabine, Busulfan, cyclophosphamide and post-transplant cyclophosphamide for a haploidentical donor transplant
Period: Overall Study
Arm/Group | Haploidentical Transplant
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.75 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Graft Rejection for Patients at Day 100
Description: Number of patients who experienced graft rejection by Day 100
Time Frame: Day 100
Population: 20 patients were treated and able to be analyzed for graft rejection
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 20
participants | 0

2. Primary Outcome: Number of Patients Who Experienced Severe Graft-versus-host Disease (GVHD)(Grade 3 or 4)
Description: Number of patients who experienced post-transplant complication (GVHD) as seen by clinical evidence
Time Frame: Day 100
Population: 17 patients were alive at Day 100 and eligible to be evaluated for grade 3-4 graft versus host disease
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 17
participants | 2

3. Secondary Outcome: Overall Survival at Day 100
Description: Overall survival is assessed, without regard to disease status, post-transplant, at Day 100.
Time Frame: Day 100
Population: 20 patients received a haploidentical transplant and therefore are eligible to be evaluated for Day 100 survival
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 20
participants | 17

4. Secondary Outcome: Non-relapse Mortality at 1 Year After Peripheral Blood Stem Cell Transplantation (PBSCT)
Description: Non-relapse mortality refers to whether a patient dies of causes related to something other than the primary disease.
Time Frame: 1 year
Population: 6 patients died prior to one year and therefore are eligible to be evaluated for non-relapse mortality.
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 6
participants | 2

5. Secondary Outcome: Achievement of >90% (Full) Donor Chimerism in the T-Cell Lineage as Measured by PCR at Day 30 Post-transplantation
Description: Chimerism analysis of peripheral blood mononuclear cells using PCR (polymerase chain reaction) for STR/VNTR (short tandme repeat/variable number tandem repeat) will be performed post transplant. On each occasion, the peripheral blood will be separated into the T-cell component (using e.g. CD3 selection) and the myeloid component (using e.g.CD14/15 selection) before assessment of chimerism.
Time Frame: Day 30
Population: 18 patients had Day 30 chimerism drawn
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 18
participants | 18

6. Secondary Outcome: Non-relapse Mortality at Day 100 After Peripheral Blood Stem Cell Transplantation (PBSCT)
Time Frame: Day 100
Population: 2 patients died before Day 100 and therefore are eligible to be evaluated for non-relapse mortality
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 2
participants | 2

7. Secondary Outcome: Achievement of >90% (Full) Donor Chimerism in the T-Cell Lineage as Measured by PCR at Day 60 Post-transplantation
Description: Chimerism analysis of peripheral blood mononuclear cells using PCR for STR/VNTR will be performed post transplant. On each occasion, the peripheral blood will be separated into the T-cell component (using e.g. CD3 selection) and the myeloid component (using e.g.CD14/15 selection) before assessment of chimerism.
Time Frame: Day 60
Population: 18 patients had chimerism drawn at Day 60
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 18
participants | 18

8. Secondary Outcome: Achievement of >90% (Full) Donor Chimerism in the T-Cell Lineage as Measured by PCR at Day 90 Post-transplantation
Description: as for outcome 7
Time Frame: Day 90
Population: 13 patients had chimerism drawn at Day 90
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 13
participants | 13

9. Secondary Outcome: Overall Survival at 12 Months
Description: Overall survival, defined as a patient being alive after transplant, is without regard to disease status.
Time Frame: 12 months
Population: 20 patients received haploidentical transplant and therefore were eligible to be evaluated for overall survival at 1 year
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 20
participants | 14

10. Secondary Outcome: Disease Free Survival at 12 Months
Description: Disease free survival refers to patients with no evidence of disease after transplant, at the 12 month time point.
Time Frame: 12 months
Population: 14 patients were alive at one year and therefore were eligible to be evaluated for disease free survival at 1 year
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 14
participants | 7

11. Secondary Outcome: Disease Free Survival at Day 100
Description: Disease free survival refers to patients with no evidence of disease after transplant, at the Day 100 time point.
Time Frame: Day 100
Population: 17 patients were alive at Day 100 and therefore were eligible to be evaluated for disease free survival at D100
Measure: Number; unit: participants
Arm/Group | Haploidentical Transplant
Number analyzed (Participants) | 17
participants | 16

ADVERSE EVENTS:
Description: Adverse Events (AEs) regardless of grade were recorded for 6mo post-transplant. Serious Adverse Events (SAEs) were reported within 24hrs of notification. Patients with baseline AE that did not experience an increase in grade (remained the same grade or lesser)were not included in the totals.
Arm/Group | Haploidentical Transplant
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical Transplant (N=20)
Acute graft versus host disease (Immune system disorders) | 1 (1) — Acute graft versus host disease as it relates to SAE reporting rather than the total number of patients who had GVHD
Ascites (Gastrointestinal disorders) | 1 (1)
BK virus (Infections and infestations) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Confusion (Nervous system disorders) | 1 (1)
Death (General disorders) | 2 (2) — This event is death as it relates to being a serious adverse event (rather than all deaths for the study)
Hemorrhagic Cystitis (Renal and urinary disorders) | 1 (1)
Hypoglycemia induced hemiparesis (Nervous system disorders) | 1 (1)
Infection with normal ANC (Infections and infestations) | 1 (1)
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia (Infections and infestations) | 2 (2)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical Transplant (N=20)
Constitutional - feeling cold (General disorders) | 2 (2)
abdominal cramping (Gastrointestinal disorders) | 10 (10)
abdominal distension (Gastrointestinal disorders) | 6 (6)
abdominal pain (Gastrointestinal disorders) | 9 (9)
abdominal tenderness (Gastrointestinal disorders) | 3 (3)
abnormal taste (Gastrointestinal disorders) | 2 (2)
agitation (Nervous system disorders) | 6 (6)
ALK PHOS (Metabolism and nutrition disorders) | 2 (2)
ALT (Hepatobiliary disorders) | 17 (17)
Altered taste (Gastrointestinal disorders) | 2 (2)
Alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ANC (Blood and lymphatic system disorders) | 17 (17)
Anemia (Blood and lymphatic system disorders) | 18 (18)
Anorexia/decreased appetite (Metabolism and nutrition disorders) | 17 (17)
Anxiety (Psychiatric disorders) | 16 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 2 (2)
AST (Hepatobiliary disorders) | 12 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7)
BK virus (Infections and infestations) | 15 (15)
Bladder pain (Renal and urinary disorders) | 5 (5)
Bladder pressure (Renal and urinary disorders) | 4 (4)
bladder spasms (Renal and urinary disorders) | 7 (7)
bloating (Gastrointestinal disorders) | 2 (2)
bradycardia (Cardiac disorders) | 2 (2)
bruising (Skin and subcutaneous tissue disorders) | 3 (3)
c-diff (Infections and infestations) | 7 (7)
cardiomyopathy (Cardiac disorders) | 3 (3)
chills (General disorders) | 15 (15)
CMV (Infections and infestations) | 11 (11)
Coag Neg Staph (Infections and infestations) | 2 (2)
confusion (Psychiatric disorders) | 6 (6)
constipation (Gastrointestinal disorders) | 8 (8)
cough (Respiratory, thoracic and mediastinal disorders) | 17 (17)
creatinine (Renal and urinary disorders) | 14 (14)
cvc bleeding (Skin and subcutaneous tissue disorders) | 2 (2)
cvc erythema (Skin and subcutaneous tissue disorders) | 4 (4)
cvc tenderness/pain (Skin and subcutaneous tissue disorders) | 4 (4)
decreased EF (Cardiac disorders) | 2 (2)
depression (Psychiatric disorders) | 13 (13)
diaphoresis (Skin and subcutaneous tissue disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 19 (19)
difficulty swallowing (Gastrointestinal disorders) | 3 (3)
dizziness (General disorders) | 5 (5)
drowsiness (General disorders) | 5 (5)
dry eyes (Eye disorders) | 2 (2)
dry lips (Skin and subcutaneous tissue disorders) | 3 (3)
dry mouth (Gastrointestinal disorders) | 5 (5)
dry skin (Skin and subcutaneous tissue disorders) | 9 (9)
edema (Blood and lymphatic system disorders) | 5 (5)
epistaxis (General disorders) | 4 (4)
erythema (Skin and subcutaneous tissue disorders) | 3 (3)
esophagitis (Gastrointestinal disorders) | 5 (5)
facial edema (Skin and subcutaneous tissue disorders) | 3 (3)
fatigue (General disorders) | 19 (19)
fever (General disorders) | 18 (18)
flat affect (Psychiatric disorders) | 4 (4)
flatulence (Gastrointestinal disorders) | 5 (5)
fluid overload (Blood and lymphatic system disorders) | 6 (6)
general deconditioning (General disorders) | 4 (4)
GERD/dyspepsia (Gastrointestinal disorders) | 14 (14)
GI distress (Gastrointestinal disorders) | 3 (3)
gram + bacteremia (Infections and infestations) | 2 (2)
hallucinations (Psychiatric disorders) | 2 (2)
headache (General disorders) | 7 (7)
hearing loss (Ear and labyrinth disorders) | 2 (2)
hematuria (Renal and urinary disorders) | 10 (10)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
hemorrhagic cystitis (Renal and urinary disorders) | 4 (4)
hemorrhoids (Skin and subcutaneous tissue disorders) | 2 (2)
hiccoughs (General disorders) | 2 (2)
hives (Immune system disorders) | 2 (2)
hyperbilirubinemia (Hepatobiliary disorders) | 8 (8)
hypercalcemia (Investigations) | 11 (20)
hyperglycemia (Investigations) | 19 (20)
hyperkalemia (Blood and lymphatic system disorders) | 12 (12)
hypermagnesemia (Blood and lymphatic system disorders) | 2 (2)
hypernatremia (Blood and lymphatic system disorders) | 9 (9)
hyperphosphatemia (Investigations) | 3 (3)
hyperpigmented skin (Skin and subcutaneous tissue disorders) | 7 (7)
hypertension (Cardiac disorders) | 11 (11)
hypoalbuminemia (Investigations) | 15 (15)
hypocalcemia (Investigations) | 14 (14)
hypoglycemia (Investigations) | 4 (4)
hypokalemia (Investigations) | 15 (15)
hypomagnesemia (Investigations) | 18 (18)
hyponatremia (Investigations) | 12 (12)
hypophosphatemia (Investigations) | 4 (4)
hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
hypotension (Cardiac disorders) | 8 (8)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
increased oral secretions (Gastrointestinal disorders) | 2 (2)
increased PT (Blood and lymphatic system disorders) | 2 (2)
insomnia (General disorders) | 14 (14)
lethargy (General disorders) | 6 (6)
lip lesion (Skin and subcutaneous tissue disorders) | 2 (2)
LE edema (Blood and lymphatic system disorders) | 10 (10)
MRSE (Infections and infestations) | 2 (2)
mucositis (Gastrointestinal disorders) | 20 (20)
myalgia (Musculoskeletal and connective tissue disorders) | 8 (8)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
nausea (Gastrointestinal disorders) | 19 (19)
neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
neck stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
neutropenic fever (General disorders) | 6 (6)
night sweats (General disorders) | 4 (4)
pain (General disorders) | 5 (5)
parainfluenza (Infections and infestations) | 5 (5)
penile pain (Reproductive system and breast disorders) | 3 (3)
periorbital edema (Eye disorders) | 2 (2)
peripheral neuropathy (Nervous system disorders) | 9 (9)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
pruritis (Skin and subcutaneous tissue disorders) | 18 (18)
pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 15 (15)
reactive airway disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
rectal discomfort (Gastrointestinal disorders) | 3 (3)
renal insufficiency (Renal and urinary disorders) | 5 (5)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
restlessness (General disorders) | 3 (3)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
rigors (General disorders) | 2 (2)
RSV (Infections and infestations) | 2 (2)
seasonal allergies (Immune system disorders) | 3 (3)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 9 (9)
shoulder discomfort (Musculoskeletal and connective tissue disorders) | 2 (2)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
sinus drainage (Respiratory, thoracic and mediastinal disorders) | 3 (3)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
skin discoloration (Skin and subcutaneous tissue disorders) | 2 (2)
skin tear (Skin and subcutaneous tissue disorders) | 2 (2)
sore throat (Gastrointestinal disorders) | 7 (7)
staph epi (Infections and infestations) | 4 (4)
stool incontinence (Gastrointestinal disorders) | 5 (5)
suprapubic pain (General disorders) | 3 (3)
tachycardia (Cardiac disorders) | 19 (19)
tachypnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
throat pain (Gastrointestinal disorders) | 4 (4)
thrombocytopenia (Blood and lymphatic system disorders) | 17 (17)
thrush (Infections and infestations) | 2 (2)
tremors (Nervous system disorders) | 4 (4)
unsteady gait (General disorders) | 2 (2)
urinary burning (Renal and urinary disorders) | 3 (3)
urinary frequency (Renal and urinary disorders) | 9 (9)
urinary incontinence (Renal and urinary disorders) | 3 (3)
urinary urgency (Renal and urinary disorders) | 5 (5)
vaginal spotting/bleeding (Reproductive system and breast disorders) | 3 (3)
visual changes (Eye disorders) | 2 (2)
vomitting (Gastrointestinal disorders) | 19 (19)
VRE (Infections and infestations) | 4 (4)
Decreased WBC (Blood and lymphatic system disorders) | 18 (18)
weakness (General disorders) | 9 (9)
weight gain (General disorders) | 2 (2)
weight loss (General disorders) | 3 (3)
wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less